# Efficacy of Intercostal CryoAnalgesia in Patients Undergoing Robot Assisted Anatomic Lung Resection

# **PROTOCOL SUMMARY**

Synopsis

| Synopsis | |
|---|---|
| Title: | Efficacy of Intercostal CryoAnalgesia in Patients Undergoing Robot |
| Chart Title: | Assisted Anatomic Lung Resection |
| Short Title: | CryoNB in Robotic Lung Resection |
| Study Design: | Prospective randomized study |
| Study Objectives: | The objectives are to determine if the addition of Cryo Nerve Block at the |
| | time of robot assisted thoracoscopic lung resection surgery will: |
| | Allow for improved postoperative analgesia as measured using |
| | Visual Analogue Scale (VAS) pain scores |
| | Allow for decreased post-operative pain medication (opioid) use |
| | Allow for accelerated recovery as measured by patient reported |
| | M.D. Anderson Symptom Inventory (MDASI) Questionnaire |
| | Increases the risk for development of neurogenic pain as |
| | measured by the Leeds Assessment of Neuropathic Symptoms |
| | and Signs (LANSS) pain scale |
| Number of Subjects: | 40 (20 in each group) |
| Sites: | Single site – Froedtert Hospital/Medical College of Wisconsin |
| | Single surgeon – Mario Gasparri, MD |
| Study Population: | Patients undergoing robot assisted thoracoscopic anatomic lung |
| | resection (pneumonectomy, bilobectomy, lobectomy or segmentectomy) |
| Inclusion Criteria: | Age 18 - 85 years male or female |
| | Acceptable surgical candidate |
| | Willing and able to return for scheduled follow-up visits |
| Exclusion Criteria: | Patients undergoing or requiring conversion to thoracotomy |
| | Patients with chronic pain syndromes requiring treatment within |
| | the last year |
| | Patients with a history of illicit drug use |
| | Patients with a history of heavy alcohol use in the last five years |
| | as determined by the principal investigator |
| | Patients currently using opioids |
| Participant Duration: | Six months |
| Study Endpoints: | Primary endpoints |
| | Visual Analogue Scale (VAS) Pain score on post-operative days |
| | 1-14, Day 30, Day 60, Day 90, Day 120, Day 150, Day 180 (or |
| | until a score of 0). |
| Pain medication use daily for 21 days post-operatively | |
| | Secondary endpoints |
| | M.D. Anderson Symptom Inventory Questionnaire on post- |
| | operative Day 1, Day 7, Day 14, Day 21, Day 30, Day 35, and |
| | Day 42 |
| | Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) |
| | score at Post-Operative Day 30, Day 90, and Day 180 |



#### Outcome measures

- VAS pain scores daily x 14 days then monthly x 6 months (or until score of 0)
- Pain medication (opioid) usage daily x 21 days
- MDASI questionnaire on POD 1 then weekly x 6 weeks
- LANSS score at 1 month, 3 months, 6 months

#### **HYPOTHESIS**

The addition of Cryo Nerve Block to a standard postoperative pain regimen will improve analgesia and facilitate recovery following robot assisted thoracoscopic anatomic lung resection

#### SPECIFIC AIMS

This study will determine if the addition of Cryo Nerve Block during robot assisted thoracoscopic anatomic lung resection surgery will:

#### **PRIMARY ENDPOINTS:**

- Allow for improved postoperative analgesia as measured using Visual Analogue Scale (VAS) pain scores
- Allow for decreased post-operative pain medication (opioid) usage

#### **SECONDARY ENDPOINTS:**

- Allow for accelerated recovery as measured by patient reported M.D. Anderson Symptom Inventory (MDASI) Questionnaire
- Increases the risk for development of neurogenic pain as measured by the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale

#### RATIONALE FOR THE PROJECT

Thoracic surgical procedures are consistently reported to be among the most painful surgical incisions currently used.<sup>1</sup> Trauma to the skin, muscle, intercostal nerves, bones and pleura all contribute and lead to activation of various pain pathways including somatic, visceral, neurogenic and phrenic.<sup>1</sup> In the short term, this pain leads to ineffective cough and pulmonary hygiene resulting in respiratory complications and prolonged hospital stays while in the longer term it leads to prolonged recovery, delayed return to work and in some instances, chronic post thoracotomy pain syndromes.<sup>2</sup> Minimally invasive approaches such as standard thoracoscopy or robotic assisted thoracoscopy have certainly decreased some of this trauma as evidenced by decreased length of stays and decreased complication rates however even with these minimally invasive techniques, recovery to 80% of baseline is 25 days<sup>3</sup> and 9.4% of patients are still using narcotics after 90-180 days.<sup>4</sup>

Several options are available in the management of pain following thoracic surgery with a multimodal pain medicine approach being most common. Opioids, unfortunately, are a relatively large part of this approach and are often relied upon despite their relatively unfavorable adverse event profile and risk for addiction. Many of the other pain adjuncts often used with thoracotomies such as epidural catheters or intraoperatively placed pain catheters are not really reasonable when using minimally invasive approaches as the hospital length of stay is 1-2 days. Intercostal cryoanalgesia has been shown to be a safe and effective strategy for post-operative pain management in patients undergoing thoracotomy. Recent studies have demonstrated the beneficial effect of cryoanalgesia for post-thoracotomy pain in reduction of opioid requirement, reduction in post-operative pain scores, and superior pulmonary function (higher FEV1 and FVC values) and that it can produce temporary neurolysis for up to two months without long-term histological nerve damage. To date it has not been studied when using minimally invasive techniques whether it be standard thoracoscopy or robotic assisted thoracoscopy but it would stand to reason that it would be equally or maybe more effective in this patient population and truly maximize the benefits of a minimally invasive approach.

We therefore propose to assess whether intra-operative intercostal cryoanalgesia using the cryoICE® probe provides superior post-operative analgesia as compared to our current standard pain management strategy in patients undergoing robotic assisted thoracoscopic anatomic lung resection and allows for decreased opioid use and more rapid recovery.

# PROJECT DESIGN AND PROTOCOL DESIGN

This is a single center, single surgeon, prospective, randomized trial examining the addition of Cryo Nerve Block during robot assisted thoracoscopic anatomic lung resection surgery

#### SUBJECTS IN THE STUDY

40 total subjects will be enrolled in the study – 20 in each group

#### **Inclusion Criteria**

- Patients undergoing robot assisted thoracoscopic anatomic lung resection surgery
- Male or female age 18 or older
- Acceptable surgical candidate
- Willing and able to return for scheduled follow-up visits

#### **Exclusion Criteria**

- Patients undergoing or requiring conversion to thoracotomy
- Patients with chronic pain syndromes requiring treatment in the last year
- Patients with a history of illicit drug use
- Patients with a history of heavy alcohol use in the last five years as determined by the principal investigator
- Patients currently using opioids

#### **CONSENT**

All patients eligible for this study will be approached for consent to enter the study in compliance with Human Research Review Committee (HRRC) standards. Consent will be obtained by the principal investigator or authorized delegate.

#### **RANDOMIZATION PROCESS**

Following the attainment of consent to enter the study, patients will be randomized to either the standard postoperative pain regimen or the standard postoperative pain regimen plus cryo nerve block by a blinded procedure where a card indicating either group will be drawn in a witnessed setting by a noninvestigator.

#### **PROCEDURE**

All patients will be assessed at baseline and then taken to the operating room for robot assisted thoracoscopic anatomic lung resection surgery. Each operation will be performed by the same surgeon and port placement will be identical (aside from laterality) in each patient. All patients will have the first two ports placed at which time an intercostal nerve block of nerves 4-9 will be performed using 0.5% Marcaine with Epinephrine. Additionally, in the study group, Cryo Nerve Block of nerves 4-9 will also be performed. To perform the cryo nerve block the 18 inch Atricure® cryoSPHERE Probe will be used in each case. The remaining ports will then be placed, the robot docked, and the procedure performed. Following the procedure, a chest tube will be placed through the camera port. Postoperatively, all patients will receive the standard post-operative pain regimen currently used by the Thoracic Surgery Service at Froedtert Hospital/Medical College of Wisconsin which consists of Tylenol and Robaxin around the clock and Ultram as first line analgesia for breakthrough pain and Oxycodone as the second line agent if necessary.

#### **RISKS AND PRECAUTIONS**

The pain management strategy outlined above, whether with or without cryo nerve block, is the current standard pain management strategy following robot assisted thoracoscopic lung

resection surgery at Froedtert Hospital/Medical College of Wisconsin. Both are routinely employed and it must be stressed that neither arm is experimental in any way with both modalities currently in use and being used successfully. What is unclear at present is which approach offers greater advantage to the patient in terms of improved analgesia and facilitation of recovery.

Risks inherent to this study are those associated with the operative procedure of robot assisted thoracoscopic lung resection surgery. To date there have been no reports of acute adverse events with cryo nerve block.

#### **DATA COLLECTED**

As shown in the schema, the following data will be collected

Preoperatively – within 30 days of surgery

- Characteristics (Age, gender, race, marital status, ECOG function, height, weight, BMI, tobacco use, major comorbidities)
- Baseline VAS Score
- Baseline MDASI
- Baseline LANSS

Intraoperatively – at time of surgery

- Procedure
- Procedure duration
- Port placement
- Intraoperative complications
- Estimated blood loss (EBL)

Postoperatively – at designated time points

- Length of stay
- Chest tube duration
- Complications
- VAS pain scores daily on post-operative Days 1-14, Day 30, Day 60, Day 90, Day 120, Day 150, Day 180 (or until score of 0).
- Pain med usage daily for post-operative Days 1-21
- MDASI questionnaire on post-operative Day 1, Day 7, Day 14, Day 21, Day 30, Day 35, and Day 42
- LANSS score at at Day 30, Day 90 and Day 180

A time frame of data collection points is shown below and the VAS scale, MDASI Questionnaire, and LANSS pain scale are included in the appendix.

| Day | Characteristics | VAS | MDASI | LANSS | Pain meds |
|----------|-----------------|-----|-------|-------|-----------|
| Baseline | Х | Χ | Х | Χ | Х |
| 0 | | | | | |
| 1 | | Χ | Х | | Х |
| 2 | | Χ | | | Х |
| 3 | | Χ | | | Х |
| 4 | | Χ | | | Χ |

| 5 | Χ | | | Χ |
|------------------|---|---|---|---|
| 6 | Χ | | | X |
| 7 | Χ | Х | | X |
| 8 | Χ | | | X |
| 9 | Χ | | | Х |
| 10 | Χ | | | X |
| 11 | Χ | | | X |
| 12 | Χ | | | X |
| 13 | Χ | | | X |
| 14 | Χ | X | | X |
| 15 | | | | X |
| 16 | | | | X |
| 17 | | | | Χ |
| 18 | | | | X |
| 19 | | | | X |
| 20 | | | | X |
| 21 | | Х | | X |
| 22 | | | | X |
| 30 (+/- 2 days) | Χ | Х | Х | |
| 35 (+/- 2 days) | | X | | |
| 42 (+/- 2 days) | | X | | |
| 60 (+/- 5 days) | Χ | | | |
| 90 (+/- 5 days) | Χ | | X | |
| 120 (+/- 5 days) | Χ | | | |
| 150 (+/- 5 days) | Χ | | | |
| 180 (+/- 5 days) | Χ | | Х | |

#### REFERENCES

- 1. Marshall K, McLaughlin K. Pain Management in Thoracic Surgery. Thorac Surg Clin 2020;30(3):339-346
- 2. Niraj G, Kelkar A, Kaushik V, et al. Audit of postoperative pain management after open thoracotomy and the incidence of chronic postthoracotomy pain in more than 500 patients at a tertiary center. J Clin Anes 2017;36:174-177
- 3. Fagundes CP, Shi Q, Vaporciyan AA, et al. Symptom recovery after thoracic surgery: Measuring patient-reported outcomes with the MD Anderson Symptom Inventory. J Thorac Cardiovasc Surg 2015;150:613-9
- 4. Brescia AA, Harrington CA, Mazurek AA, et al. Factors associated with new persistent opioid usage after lung resection. Ann Thorac Surg 2019;107(2):363–868

5. Sepsas E, Misthos P, Anagnostopulu M, et al. The role of intercostal cryoanalgesia in post-thoracotomy analgesia. Interact Cardiovasc Thorac Surg 2013;16:814-818

6. Moorjani N, Zhao F, Tian Y, et al. Effects of cryoanalgesia on post-thoracotomy pain and on the structure of intercostal nerves: a human prospective randomized trial and a histological study. Eur J Cardiothorac Surg 2001;20:502-507.

# **APPENDIX I - Eastern Cooperative Oncology Group (ECOG) Performance Status**

| GRADE | ECOG PERFORMANCE STATUS |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry |
| | out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all selfcare but unable to carry out any work |
| | activities; up and about more than 50% of waking hours |
| 3 | Capable of only limited selfcare; confined to bed or chair more than 50% of |
| | waking hours |
| 4 | Completely disabled; cannot carry on any selfcare; totally confined to bed or |
| | chair |
| 5 | Dead |

### **APPENDIX II - Visual Analogue Scale Pain Score**

# UNIVERSAL PAIN ASSESSMENT TOOL

This pain assessment tool is intended to help patient care providers assess pain according to individual patient needs.

Explain and use 0-10 Scale for patient self-assessment. Use the faces or behavioral observations to interpret expressed pain when patient cannot communicate his/her pain intensity.



### Appendix III - MD Anderson Symptom Inventory (MDASI) Questionnaire

# M. D. Anderson Symptom Inventory (MDASI) Core Items

Part I. How severe are your symptoms?

People with cancer frequently have symptoms that are caused by their disease or by their treatment. We ask you to rate how severe the following symptoms have been *in the last 24 hours*. Please fill in the circle below from 0 (symptom has not been present) to 10 (the symptom was as bad as you can imagine it could be) for each item.

| | | Not<br>Present | SC 2-8 7 | 0.000 | | 9 8 7 | 0.102.1 | | D- 81 | 107-0-2 | 0.000 | Bad As You<br>Imagine |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | . 3 | 4 | 5 | : 6 | 7 | ; 8 | 9 | : 10 |
| 1. | Your pain at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 2 | Your fatigue (tiredness) at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 3. | Your nausea at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 4 | Your disturbed sleep at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 5. | Your feelings of being distressed (upset) at its WORST | , 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 6. | Your shortness of breath at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 7. | Your problem with remembering things at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 8. | Your problem with lack of appetit<br>at its WORST? | ° 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 9. | Your feeling drowsy (sleepy) at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 10 | Your having a dry mouth at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 11. | Your feeling sad at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 12. | Your vomiting at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| 13. | Your numbness or tingling at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

# Appendix IV – Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scale

| | In the area where you have pain, do you also have "pins and needles", tingling or prickling sensations? | |
|---|---|---|
| | NO − I don't get these sensations | 0 |
| | YES – I get these sensations | 5 |
| 2 | Does the painful area change colour (perhaps look mottled or more red) when the pain is particularly bad? | |
| | □ NO – The pain does not affect the colour of my skin | 0 |
| | YES – I have noticed that the pain does make my skin look different from normal. | 5 |
| | Does your pain make the affected skin abnormally sensitive to touch? Getting unpleasant sensations or pain when lightly stroking the skin might describe this. | |
| | NO – The pain does not make my skin abnormally sensitive to touch. | 0 |
| | YES – My skin in that area is particularly sensitive to touch. | 3 |
| | Does your pain come on suddenly and in bursts for no apparent reason when you are completely still? Words like "electric shocks", jumping and bursting might describe this. | |
| | □ NO – My pain doesn't really feel like this. | 0 |
| | ☐ YES – I get these sensations often. | 2 |
| | In the area where you have pain, does your skin feel unusually hot like a burning pain? | |
| | NO − I don't have burning pain | 0 |
| | YES – I get burning pain often | 1 |
| 6. | Gently rub the painful area with your index finger and then rub a non-painful area (for example, an area of skin further away or on the opposite side from the painful area). How does this rubbing feel in the painful area? | |
| | ☐ The painful area feels no different from the non-painful area | 0 |
| | ☐ I feel discomfort, like pins and needles, tingling or burning in the painful area that is different from the non-painful area. | 5 |
| | Gently press on the painful area with your finger tip and then gently press in the same way onto<br>a non-painful area (the same non-painful area that you chose in the last question). How does this<br>feel in the painful area? | |
| | The painful area does not feel different from the non-painful area. | 0 |
| | ☐ I feel numbness or tenderness in the painful area that is different from the non-painful area. | 3 |
| | Total score: | |
| | Scoring a score of 12 or more suggests pain of predominantly neuropathic origin | |